CLINICAL TRIAL: NCT03917992
Title: The Baseline Features and CHA2DS2 VASc /HAS BLED Scores of Jordanian Patients With Atrial Fibrillation and the One Year Outcome
Brief Title: The Jordan Atrial Fibrillation Study: Baseline Risk Scores and One Year Outcome
Status: Completed | Type: Observational
Sponsor: Ayman J Hammoudeh, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Ayman J Hammoudeh, MD, FACC, The Jordanian Comprehensive Center For Electophysiologic Heart Disease, Jordan Collaborating Cardiology Group
Organization: Jordan Collaborating Cardiology Group (Other)
Other Study IDs: JOAF1Y
Record Dates: First submitted 2019-04-14; First posted 2019-04-17 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Jordanian AF study, the first of its kind in Jordan, will evaluate patients with AF in an in-patient and out-patient settings. The morbidity and mortality associated with AF has not been studied in this region especially with the relation to the HAD BLED and CHADS VAC score.

DETAILED DESCRIPTION:
The investigators are introducing The Jordan Atrial Fibrillation Study: Baseline Risk Scores and One Year Outcome" which is an investigator initiated, prospective, non interventional, observational study.

Medical research and clinical studies in Jordan are two basic responsibilities of all medical sectors in the country. Despite the drastic growth and advances of the medical services, the volume of the local medical research is, at best estimate, scarce. The emerging role of private medical groups, in cooperation with other medical sectors and medical schools, in conducting, presenting, and publishing such studies should be encouraged and welcomed by the other medical sectors in the country. A major indicator of judging the credibility and quality of any medical research project is to look at the conferences the research was presented at and the journals it was published in.

This is the 9th major project of the Jordan Collaborating Cardiology Group (JCC) in collaboration with the Jordan AF Study Group. (see Appendix 2. Timeline of our studies) The first project was JoHARTS (1-5) that evaluated coronary risk factors and dyslipidemia in 5000 individuals with ACS, stable CAD, and non CAD patients. The 2nd project was CAPRIS (6,7) evaluated the prognostic implications of hs-CRP in ACS from admission to 1 year. The 3rd project was MINTOR that evaluated onset, triggers, reperfusion strategies and hospital mortality in more than 950 Jordanians with acute ST elevation MI (8-10). The 4th project was GLORY study that evaluated the prevalence of glucometabolic states among ACS patients, prognosis up to 1 year, and TIMI risk score (11-15). The 5th was JoPCR1 that evaluated outcome post PCI in 2426 ACS and non ACS patients in 12 tertiary care centers for the incidence of death, stent thrombosis, revascularization, bleeding, impact of gender, DM, renal dysfunction and age on outcome, GRACE and CRUSADE risk scores (16-18). The 6th is the colchicine study of AF prevention in open heart surgery, one is completed with 1 mg dose and one is ongoing with reduced dose (19). The 7th and 8th projects are ongoing and study statin eligibility in patients admitted with MI (Statin EPIC) and decade or more survivors after coronary revascularization.

The Jordanian AF study, the first of its kind in Jordan, will evaluate patients with AF in an in-patient and out-patient settings.

Study Objectives

1. To study the demographic baseline features of AF patients, risk factors, and comorbid diseases, and types of AF.
2. To study CHADS2 VA2Sc score and HAS BLED scores in these patients.
3. To study patterns of treatment of AF, especially the use of oral anticoagulation and concomitant antiplatelet therapy.
4. To study 1 year incidence of stroke and systemic embolization and other cardiovascular events up to one year of follow up.
5. To present these findings in regional and international conferences and publish them.

The study PI is Dr Nazih Kadri. The assistant to the PI is Dr Eisa Ghanma. The director of the proceedings is Dr A Hammoudeh, and the assistant to the study director, Dr Ahmad Tamari will aid in study clinical initiation, clinical form development, analysis of data and manuscript writing along with the whole team of PI, Co PI, study director and other investigators.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Admission with atrial fibrillation or clinic visit for atrial fibrillation
* Signing the consent form

Exclusion Criteria:

* Age less than 18 years
* Refusal of signing the censent form
* Grave systemic disease with high probability of in hospital death

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive admissions aged 18+ years with new onset or known AF Admitted to participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 2020 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Stroke and systemic embolization at one year | one year
  Stroke that develops from enrollment to one year of follow up (Scale: 0= no stroke at one year, 1= stroke at one year). Systemic embolization that develops in any arterial bed other than the brain from enrollment to one year of follow up (Scale: no systemic embolization at one year =0, systemic embolization at one year=1)
Major bleeding events at one year | one year
  Major bleeding events from enrollment to one year of follow up including: intracranial bleeding (scale: present= 1, absent=0), hospitalization for bleeding (scale: present=1, absent=2), hemoglobin decrease more than 2 gm/dL (scale: 1=present, 2=absent), and /or transfusion (scale: 1=present, 0=absent).

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Hammoudeh, MD, FACC, Study Chair — Cardiology Dept, Istishari Hospital, Amman, Jordan
Locations (8):
- Jordan (8):
  - Istishari Hospital, Amman
  - The University of Jordan, Amman
  - Ep Clinics Khalidi S, Amman
  - Integrated Center for Cardiovascular and Electric Diseases, Amman
  - Jordan Hospital, Amman
  - Khalidi Hospital & Medical Center, Amman
  - Specialty Hospital, Amman
  - King Abdullah University Hospital, Irbid

IPD SHARING:
Plan to Share IPD: Undecided
We will make available to researchers the clinical from of the study and eventually the results and publications

REFERENCES:
- [Derived] Abdin B, Abuqweider E, Alhaddad I, Shabaneh R, Bader G, Bader T, Abu-Shaban M, Salah Q, Hammoudeh A. The Effect of Multimorbidity and Anticoagulation Use in Patients with Atrial Fibrillation on The One-Year Outcome: Analysis from Jordan Atrial Fibrillation (JoFIB) Study - A Prospective Cohort Study. BMJ Open. 2025 Dec 28;15(12):e102661. doi: 10.1136/bmjopen-2025-102661. PMID 41461398
- [Derived] Hammoudeh A, Badaineh Y, Tabbalat R, Ahmad A, Bahhour M, Ja'ara D, Shehadeh J, Jum'ah MA, Migdad A, Hani M, Alhaddad IA. The Intersection of Atrial Fibrillation and Coronary Artery Disease in Middle Eastern Patients. Analysis from the Jordan Atrial Fibrillation Study. Glob Heart. 2024 Mar 12;19(1):29. doi: 10.5334/gh.1312. eCollection 2024. PMID 38505303
- [Derived] Alrabadi N, Al-Nusair M, Haddad R, Alburie L, Mhaidat N, Aljarrah M, Hamoudeh A. Cardiovascular medications used for comorbid diseases in patients with atrial fibrillation. The JoFib study. Eur J Clin Pharmacol. 2024 Apr;80(4):545-552. doi: 10.1007/s00228-024-03622-8. Epub 2024 Jan 23. PMID 38253701
- [Derived] Al-Makhamreh H, Alrabadi N, Haikal L, Krishan M, Al-Badaineh N, Odeh O, Barqawi T, Nawaiseh M, Shaban A, Abdin B, Khamies L, Hammoudeh A. Paroxysmal and Non-Paroxysmal Atrial Fibrillation in Middle Eastern Patients: Clinical Features and the Use of Medications. Analysis of the Jordan Atrial Fibrillation (JoFib) Study. Int J Environ Res Public Health. 2022 May 19;19(10):6173. doi: 10.3390/ijerph19106173. PMID 35627709
- [Derived] Alhaddad Z, Hammoudeh A, Khader Y, Alhaddad IA. Demographics and Risk Profile of Elderly Middle Eastern Patients with Atrial Fibrillation: The Jordan Atrial Fibrillation (JoFib) Study. Vasc Health Risk Manag. 2022 Apr 15;18:289-295. doi: 10.2147/VHRM.S360822. eCollection 2022. PMID 35449533
- [Derived] Hammoudeh AJ, Khader Y, Kadri N, Al-Mousa E, Badaineh Y, Habahbeh L, Tabbalat R, Janabi H, Alhaddad IA. Adherence to the 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline on the Use of Oral Anticoagulant Agents in Middle Eastern Patients with Atrial Fibrillation: The Jordan Atrial Fibrillation (JoFib) Study. Int J Vasc Med. 2021 Apr 8;2021:5515089. doi: 10.1155/2021/5515089. eCollection 2021. PMID 33898065